CLINICAL TRIAL: NCT05649657
Title: Effect of Lifestyle Intervention in Patients With Chronic Kidney Disease on Fitness and Immune Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202201244B0A3
Record Dates: First submitted 2022-11-07; First posted 2022-12-14 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2022-10

CONDITIONS: End-stage Renal Disease (ESRD)
Keywords: exercise; hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hemodialysis patients with exercise training intervention (Experimental): The participants under hemodialysis for over 3 months will go through three phases: 3-month control, 6-month intervention, and 3-month maintenance. No intervention will be performed in the control and maintenance phases
  Interventions: Other: Cyclic aerobic and resistance training

INTERVENTIONS:
Other: Cyclic aerobic and resistance training — Two options for the participants to choose from. First, a home-based program. The participant will be requested to wear a heart rate recorder during home exercise. Second, a hospital-based program. The participants visit the rehabilitation center twice weekly to receive supervised exercise therapy. The exercise prescription comprises aerobic and resistance training. The intensity is set initially at ventilatory anaerobic threshold and gradually titrated up to respiratory compensatory point based on the breath-by-breath cardiopulmonary exercise testing. The duration is 25~35 minutes per session plus a 5-minute warm-up and 5-min cool-down. The frequency is 2~3 sessions per week and about 70 sessions in total.

SUMMARY:
To assess the efficacy of a 6-month lifestyle intervention in patients with end-stage renal disease(ESRD), we plan to conduct a self-controlled clinical trial. 34 participants receiving chronic HD will be enrolled. Each participant will go through three phases: 3-month control, 6-month intervention, and 3-month maintenance. No intervention will be performed in the control and maintenance phases. The lifestyle intervention will comprise care from a multidisciplinary team, including a nephrologist, nurse practitioner, physiatrist, and dietitian. The exercise training component is an in-hospital supervised training 2~3 times weekly for 6 months. Cyclic aerobic and resistance training will be performed. Assessment will be performed every three months and 5 times in total, including cardiopulmonary exercise testing, isokinetic quadriceps strength testing, hand grip strength, body composition analysis, Chinese Kidney Disease and Quality of Life questionnaire, self-recorded physical activity, and Mini Nutritional Assessment. The aim of this study is to assess the efficacy of a lifestyle intervention in patients with chronic kidney disease (CKD) on physical fitness, quality of life, and immunity. It is hypothesized that the lifestyle intervention will elicit a significant benefit in the aforementioned parameters and will last until the maintenance phase.

DETAILED DESCRIPTION:
The prevalence of end-stage renal disease is high, especially in Taiwan. Cardiovascular diseases and infection are the major causes of morbidity. Though evidence is clear that exercise training in this population is beneficial to fitness、quality of life、morbidity, it is seriously underused. Poor physical fitness is known to associate with high-leveled systemic inflammation and immune dysregulation but the detailed relationship remains unclear in the ESRD population. Moreover, though exercise improves low physical fitness, available research concerning its effect on the pro-/anti-inflammatory immune response is scarce. Does supervised lifestyle intervention has the potential to improve physical fitness, and quality of life in patients receiving maintenance hemodialysis (HD)? To assess the efficacy of a 6-month lifestyle intervention in patients under HD, we plan to conduct a self-controlled clinical trial. No intervention will be performed in the control and maintenance phases. The lifestyle intervention will comprise care from a multidisciplinary team, including a nephrologist, nurse practitioner, physiatrist, and dietitian. The exercise training component is in-hospital supervise training 2~3 times weekly for 6 months. Cyclic aerobic and resistance training will be performed. Assessment will be performed every three months and 5 times in total, including cardiopulmonary exercise testing, isokinetic quadriceps strength testing, hand grip strength, body composition analysis, Chinese Kidney Disease and Quality of Life questionnaire, self-recorded physical activity, and Mini Nutritional Assessment. The aim of this study is to assess the efficacy of a lifestyle intervention in patients under HD on physical fitness, and quality of life. It is hypothesized that the lifestyle intervention will elicit a significant benefit in the aforementioned parameters and will last until the maintenance phase.

ELIGIBILITY:
Inclusion Criteria:

* patients who are on HD for longer than 6 months
* under the permission of their nephrologist
* adequately dialyzed (most recent Kt/V > 1.2) and stable during dialysis in the past 3 months

Exclusion Criteria:

* occurrence of hyperkalemia in the past 3 months
* comorbid medical, physical, and mental conditions that contraindicate exercise
* unstable cardiac conditions (eg, unstable angina, heart failure or symptomatic severe aortic stenosis, etc.)
* disabling orthopedic and neuromuscular diseases

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Chun Huang, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Huang SC, Fang JT, Huang YC, Lin CY, Hsiao CC. From gains to decline: effects of structured pre-dialytic exercise training and detraining on physical fitness, quality of life, and inflammation in haemodialysis patients. J Rehabil Med. 2025 Oct 22;57:jrm44067. doi: 10.2340/jrm.v57.44067. PMID 41126503

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were eligible for inclusion if they had been undergoing hemodialysis (HD) for more than 3 months, were over 20 years of age, had adequate dialysis (Kt/V > 1.2), obtained approval from their nephrologist, and were able to walk independently for more than 10 meters. Exclusion criteria included recent hyperkalemia, medical or orthopedic conditions, muscular or psychological disorders, and a history of heart failure or inability to participate in cycling or exercise testing.
Pre-assignment Details: This study employed self-controlled design. Over the study period, each participant underwent assessments at five time points (T1, T2, T3, T4, and T5) with about 3 months between each time point. Between T1 and T2 was the control phase, the participants received usual medical care only. Between T2 and T4 was the training phase, exercise training and nutrition education were implemented. The T4-T5 follow-up phase monitored changes after training cessation with standard medical care only.
Groups:
- Hemodialysis Partipants: Each participant will undergo 3-month control, 6-month intervention, and 3-month maintenance. There was no intervention in the control and maintenance phases.
Period: Overall Study
Arm/Group | Hemodialysis Partipants
Started | 34
Completed | 22
Not Completed | 12

BASELINE CHARACTERISTICS:
Groups:
- Self-controlled Study: A three-phase self-controlled design was used: 3-month control, 6-month training (72 sessions), and 3-month follow-up.
Arm/Group | Self-controlled Study
Number analyzed (Participants) | 22
Age, Continuous [Median (Inter-Quartile Range); unit: year] | 62 [52 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Taiwan | 22
peak VO2 [Median (Inter-Quartile Range); unit: ml/min/kg] | 14.8 [12.7 to 16.6]

OUTCOME MEASURES:

1. Primary Outcome: Peak Oxygen Consumption
Description: cardiopulmonary exercise testing
Time Frame: 1 year
Population: 22 completed the 72-session training at T4 and after follow-up at T5
Measure: Median (Inter-Quartile Range); unit: ml/min/kg
Groups:
- Self-controlled Study: The participants receiving maintenance hemodialysis for over 3 months went through three phases: 3-month control, 6-month intervention, and 3-month maintenance. There was no intervention in the control and maintenance phases.
Arm/Group | Self-controlled Study
Number analyzed (Participants) | 22
ml/min/kg | 3.07 [1.06 to 5.95]

2. Primary Outcome: Inflammatory Cytokines
Description: Interleukin (IL)-6 concentration was detected in plasma using the BD Cytometric Bead Array (CBA) Human Inflammatory Cytokines Kit (Becton-Dickinson) and analyzed with FCAP Array™ software .
Time Frame: 1 year
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Hemodialysis Partipants
Number analyzed (Participants) | 22
pg/ml | 2.84 [2.01 to 6.08]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Self-controlled Study
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT05649657/Prot_SAP_000.pdf